CLINICAL TRIAL: NCT05643755
Title: Investigating the Effect of Preoperative Image-based Education on Postoperative Satisfaction of Patients Undergoing First-time Dermatologic Surgery
Brief Title: Preoperative Image-based Education Effect on Postoperative Satisfaction of Patients Undergoing First-time Dermatologic Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of personnel to complete study.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00357538
Record Dates: First submitted 2022-11-30; First posted 2022-12-09 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Skin Cancer; Skin Wound
Keywords: Mohs Surgery; Wide Local Excision
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention group: educational material provided on the day of surgery containing pictographic and written education material on wound appearance following primary closure after Mohs Micrographic Surgery (MMS) or Wide Local Excision (WLE)
  Interventions: Other: Preoperative image-based education
- Control (No Intervention): Control group: standard clinical care

INTERVENTIONS:
Other: Preoperative image-based education — Intervention group: education handout containing pictographic and written education material on wound appearance following primary closure after Mohs Micrographic Surgery (MMS) or Wide Local Excision (WLE)
  Arms: Intervention

SUMMARY:
This research study aims to understand whether visual and written education on wound appearance can improve patients' experience and understanding of what their wound will look like following dermatologic surgery.

DETAILED DESCRIPTION:
Undergoing surgery is a stressful process for many patients. By its nature, dermatologic surgery carries additional stressors given that it is performed on the skin, a very cosmetically sensitive area. In our dermatologic surgery practice, we have found that patients are often surprised by the length of their surgical wound immediately post-surgery; many have expressed confusion about the length of the wound relative to the much smaller targeted lesion.

Our research study will utilize image-based education prior to patients' first dermatologic surgery to determine whether this intervention helps patients feel more satisfied with their wound appearance immediately post-surgery. Our primary hypothesis is that patients who are undergoing dermatologic surgery for the first time will benefit from image-based education about the surgical wound closure process. We hypothesize that a greater proportion of such patients would feel more satisfied and less distressed with the cosmetic outcomes immediately after their surgery relative to patients who did not receive image-based education.

If this hypothesis is found to be true, we will conclude that there is a need for better patient education prior to their dermatologic surgery procedure. We hope that this study will create a framework for sharing educational resources with patients so that they may set expectations as to surgical outcomes. These findings may also be relevant to other surgical procedures where patient satisfaction would be improved by the implementation of pre-operative education.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria: Adult patients (ages 18-100) who will be undergoing dermatology surgery at Johns Hopkins. We will include only patients who are undergoing their first dermatology surgery. Only patients whose incisions are closed with primary closure will be eligible.

Exclusion Criteria:

* Patients who have already undergone dermatology surgery.
* Patients whose incisions are not closed with primary closure

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction with wound appearance immediately after surgery in control vs. intervention groups as assessed by the Modified Skin Cancer Index questionnaire | At time of surgery
  Whether the wound appearance is as expected, worse than expected, or better than expected immediately after surgery in control vs. intervention groups. We will administer the Modified Skin Cancer Index questionnaire to determine patient satisfaction with their wound appearance and compare satisfaction between control and intervention groups.

SECONDARY OUTCOMES:
Patient factors associated with satisfaction with wound appearance as assessed by Modified Skin Cancer Index questionnaire | Up to 4 weeks after surgery
  We will collect information from the patient chart (including demographic factors, medical comorbidities, wound characteristics) to correlate these factors with patient satisfaction with their wound appearance

CONTACTS AND LOCATIONS:
Overall Officials: Elise Ng, MD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sobanko JF, Sarwer DB, Zvargulis Z, Miller CJ. Importance of physical appearance in patients with skin cancer. Dermatol Surg. 2015 Feb;41(2):183-8. doi: 10.1097/DSS.0000000000000253. PMID 25654193
- [Background] Dixon AJ, Dixon MP, Dixon JB. Prospective study of long-term patient perceptions of their skin cancer surgery. J Am Acad Dermatol. 2007 Sep;57(3):445-53. doi: 10.1016/j.jaad.2007.02.006. PMID 17707149
- [Background] Cassileth BR, Lusk EJ, Tenaglia AN. Patients' perceptions of the cosmetic impact of melanoma resection. Plast Reconstr Surg. 1983 Jan;71(1):73-5. doi: 10.1097/00006534-198301000-00016. PMID 6849025
- [Background] Long J, Rajabi-Estarabadi A, Levin A, Nami N, Nouri K. Perioperative Anxiety Associated With Mohs Micrographic Surgery: A Survey-Based Study. Dermatol Surg. 2022 Jul 1;48(7):711-715. doi: 10.1097/DSS.0000000000003455. Epub 2022 Apr 18. PMID 35438652
- [Background] Pereira L, Figueiredo-Braga M, Carvalho IP. Preoperative anxiety in ambulatory surgery: The impact of an empathic patient-centered approach on psychological and clinical outcomes. Patient Educ Couns. 2016 May;99(5):733-8. doi: 10.1016/j.pec.2015.11.016. Epub 2015 Nov 26. PMID 26654958
- [Background] Sobanko JF, Da Silva D, Chiesa Fuxench ZC, Modi B, Shin TM, Etzkorn JR, Samimi SS, Wanat KA, Miller CJ. Preoperative telephone consultation does not decrease patient anxiety before Mohs micrographic surgery. J Am Acad Dermatol. 2017 Mar;76(3):519-526. doi: 10.1016/j.jaad.2016.09.027. Epub 2016 Dec 4. PMID 27923500
- [Background] Arzeno J, Liu R, Goldbach H, Moon D, Soriano T, Beynet D, Greco J, Ms MS, Kim J. Effect of pre-operative informational video on Mohs surgery patient experience. Dermatol Online J. 2021 Jun 15;27(6). doi: 10.5070/D327654069. No abstract available. PMID 34387069
- [Background] Patel P, Malik K, Khachemoune A. Patient education in Mohs surgery: a review and critical evaluation of techniques. Arch Dermatol Res. 2021 May;313(4):217-224. doi: 10.1007/s00403-020-02119-5. Epub 2020 Aug 12. PMID 32785836